CLINICAL TRIAL: NCT00060944
Title: A Randomized, Multicenter, Open-label Study of Yondelis (ET-743 Ecteinascidin) Administered by 2 Different Schedules (Weekly for 3 of 4 Weeks vs. q3 Weeks) in Subjects With Locally Advanced or Metastatic Liposarcoma or Leiomyosarcoma Following Treatment With an Anthracycline and Ifosfamide
Brief Title: A Study to Assess Treatment With 2 Different Dosing Schedules of Trabectidin Administered to Patients With Advanced Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR004336; ET743-STS-201 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2003-05-16; First posted 2003-05-19 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-08

CONDITIONS: Liposarcoma; Leiomyosarcoma
Keywords: Trabectedin; Yondelis; ET-743; Ecteinascidin; Anthracycline; Ifosfamide; Dexamethasone; Intravenous; Cancer; Malignant; Metastatic
MeSH Terms: conditions — Liposarcoma; Leiomyosarcoma; Neoplasms; Neoplasm Metastasis | interventions — Trabectedin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yondelis weekly schedule (Experimental): Yondelis weekly schedule: 0.58 mg/m2 administered as a 3-hour i.v. infusion on Days 1 8 and 15 of each 28-day treatment cycle. Patients will be pretreated with 10 mg of dexamethasone i.v. 30 minutes prior to each infusion.
  Interventions: Drug: Yondelis; Drug: Dexamethasone
- Yondelis once every 3 weeks schedule (Experimental): Yondelis once every 3 weeks schedule: 1.5 mg/m2 administered as a 24-hour i.v. infusion on Day 1 of every 21-day treatment cycle. Patients will be pretreated with 20 mg of dexamethasone i.v. on Day 1 of each treatment cycle 30 minutes prior to each infusion.
  Interventions: Drug: Yondelis; Drug: Dexamethasone

INTERVENTIONS:
Drug: Yondelis — 1.5 mg/m2 administered as a 24-hour i.v. infusion on Day 1 of every 21-day treatment cycle.
  Arms: Yondelis once every 3 weeks schedule
Drug: Yondelis — 0.58 mg/m2 administered as a 3-hour i.v. infusion on Days 1, 8, and 15 of each 28-day treatment cycle.
  Arms: Yondelis weekly schedule
Drug: Dexamethasone — Pretreatment with 10 mg of dexamethasone i.v. 30 minutes prior to each Yondelis infusion on Days 1, 8, and 15 of each 28-day treatment cycle.
  Arms: Yondelis weekly schedule
Drug: Dexamethasone — Pretreatment with 20 mg of dexamethasone i.v. on Day 1 of each 21- day treatment cycle, 30 minutes prior to each Yondelis infusion.
  Arms: Yondelis once every 3 weeks schedule

SUMMARY:
The purpose of this study is to test the safety and effectiveness of an investigational chemotherapy agent in patients with types of advanced cancer referred to as liposarcoma or leiomyosarcoma.

DETAILED DESCRIPTION:
This is an open-label (patients will know the names of the study drugs they receive), randomized (patients will be assigned by chance to receive 1 of 2 treatment schedules with trabectidin) study designed to examine the the survival, safety, and pharmacokinetics (blood levels) trabectedin when administered to patients with 2 types of cancer (Liposarcoma or Leiomyosarcoma) who have received treatment with other anti-cancer therapy (Anthracycline and/or Ifosfamide). Trabectedin (also referred to as Yondelis) is a drug being developed to treat patients with cancer. Yondelis will be administered intravenously (i.v.) via a central catheter (tube) into a central vein once a week (0.58 mg/m2 as a 3-hour infusion on Days 1, 8, and 15 of each 28-day treatment cycle) or once every 3 weeks (1.5 mg/m2 administered as a 24-hour infusion on Day 1 of every 21-day treatment cycle) until disease progression. Patients in each arm will be pretreated with 20 mg of dexamethasone i.v. 30 minutes prior to each infusion.

ELIGIBILITY:
Inclusion Criteria:

* Have advanced liposarcoma or leiomyosarcoma that has metastasized (spread)
* Have a pathology specimen available for centralized review
* Have progressive or relapsed (reappearance of) disease, received treatment with anthracycline and/or ifosfamide before enrollment in study, and have at least one measurable tumor lesion
* Have adequate bone marrow, liver and kidney function
* Have Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Exclusion Criteria:

* Previous exposure to Yondelis i.v. formulation, ET-743 (ecteinascidin)
* Cancer that has metastasized (spread) to the central nervous system
* Active viral hepatitis or chronic liver disease
* Unstable cardiac (heart) condition including congestive heart failure or angina pectoris (heart pain), myocardial infarction (heart attack) within 1 year before enrollment
* History of another neoplastic (malignant or nonmalignant tumor) disease (except basal cell carcinoma or cervical carcinoma adequately treated), unless in remission for 5 years or more before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2003-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (39):
- United States (20):
  - Los Angeles, California
  - Aurora, Colorado
  - Coeur d'Alene, Idaho
  - Park Ridge, Illinois
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - Newark, New Jersey
  - New York, New York
  - Cleveland, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Houston, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Australia (4):
  - East Melbourne
  - Newcastle
  - Perth
  - Woodville
- Leuven, Belgium
- Canada (5):
  - Calgary, Alberta
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Edmonton
- France (2):
  - Lyon
  - Villejuif
- Düsseldorf, Germany
- Russia (4):
  - Moscow
  - Obninsk
  - Saint Petersburg
  - Samara
- Spain (2):
  - Barcelona
  - Valencia

REFERENCES:
- See also: Demetri GD et al. J Clin Oncol. 2009;27(25):4188-96. — http://www.ncbi.nlm.nih.gov/pubmed/19652065

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated the efficacy and safety of of trabectedin in participants with locally advanced or metastatic L-sarcoma whose disease had relapsed or become refractory after treatment with an anthracycline and ifosfamide. The study was conducted between 12 May 2003 and 23 April 2008 and recruited participants from 9 countries worldwide.
Pre-assignment Details: In this study 271 participants were enrolled of which 270 participants (134 in the Trabectedin 1.5 mg/m2 group and 136 in the Trabectedin 0.58 mg/m2 group) were randomized as 1 participant was enrolled twice. Of these, 260 participants were treated with trabectedin including 130 participants in each treatment group.
Groups:
- Trabectedin 1.5 mg/m2: Participants received trabectedin as a 24-hour intravenous (IV) infusion at a starting dose of 1.5 mg/m2 on Day 1 of each 21-day treatment cycle, with 20 mg dexamethasone administered IV 30 min before each trabectedin infusion.
- Trabectedin 0.58 mg/m2: Participants received trabectedin as a 3-hour intravenous (IV) infusion at a starting dose of 0.58 mg/m2 on Days 1, 8, and 15 of each 28-day treatment cycle, with 10 mg dexamethasone administered IV 30 min before each trabectedin infusion
Period: Overall Study
Arm/Group | Trabectedin 1.5 mg/m2 | Trabectedin 0.58 mg/m2
Started | 136 | 134
Treated | 130 | 130
Completed | 0 | 0
Not Completed | 136 | 134
Not completed — Adverse Event | 12 | 10
Not completed — Death | 2 | 3
Not completed — Withdrawal by Subject | 18 | 5
Not completed — Disease Progression | 93 | 94
Not completed — Lost to Follow-up | 1 | 0
Not completed — Subject Ineligible To Continue | 2 | 1
Not completed — Treatment Switch | 0 | 13
Not completed — Other | 2 | 4
Not completed — randomized but not treated | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trabectedin 1.5 mg/m2 | Trabectedin 0.58 mg/m2 | Total
Number analyzed (Participants) | 136 | 134 | 270
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (9.95) | 53.4 (10.7) | 53.1 (10.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 78 | 170
  Male | 44 | 56 | 100
Region of Enrollment [Number; unit: participants]
  Australia | 3 | 1 | 4
  Belgium | 1 | 2 | 3
  Canada | 13 | 11 | 24
  France | 5 | 12 | 17
  Germany | 2 | 0 | 2
  Italy | 5 | 3 | 8
  Russia | 15 | 13 | 28
  Spain | 3 | 0 | 3
  United States Of America | 89 | 92 | 181

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression- Independent Review
Description: Time to Progression was defined as time between randomization and the first documentation of disease progression or death due to progressive disease.
Time Frame: From randomization to the first documentation of disease progression or death due to progressive disease, whichever occurs first, assessed up to 5 years
Population: All participants who were randomly assigned to one of the two schedules, independent of whether they received trabectedin or not.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trabectedin 1.5 mg/m2 | Trabectedin 0.58 mg/m2
Number analyzed (Participants) | 136 | 134
months | 3.7 [2.1 to 5.4] | 2.3 [2.0 to 3.5]
Statistical Analysis 1: Comparison: Trabectedin 1.5 mg/m2 vs Trabectedin 0.58 mg/m2; Test type: Superiority or Other; p = 0.0302, Log Rank; Hazard Ratio (HR) = 0.734, 95% CI 2-sided [0.554 to 0.974]

2. Secondary Outcome: Percentage of Participants Objective Response - Independent Review
Description: Percentage of participants with objective response based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed CR defined as disappearance of all target lesions. Confirmed PR defined as greater than or equal to 30 percent decrease in sum of the longest dimensions (LD) of the target lesions taking as a reference the baseline sum LD according to RECIST. Confirmed responses are those that persist on repeat imaging study greater than or equal to 4 weeks after initial documentation of response.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trabectedin 1.5 mg/m2 | Trabectedin 0.58 mg/m2
Number analyzed (Participants) | 136 | 134
Percentage of participants | 5.1 [2.1 to 10.3] | 1.5 [0.2 to 5.3]

3. Secondary Outcome: Duration of Response - Independent Review
Description: Duration of response based on assessment of confirmed CR or confirmed PR according to RECIST. Confirmed CR defined as disappearance of all target lesions. Confirmed PR defined as greater than or equal to 30 percent decrease in sum of the LD of the target lesions taking as a reference the baseline sum LD according to RECIST. Confirmed responses are those that persist on repeat imaging study greater than or equal to 4 weeks after initial documentation of response. Kaplan-Meier estimation of response duration was used to account censored participants with ongoing response.
Time Frame: as for outcome 1
Population: All participants who were randomly assigned to one of the two schedules, independent of whether they received trabectedin or not. Participants with confirmed response only were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trabectedin 1.5 mg/m2 | Trabectedin 0.58 mg/m2
Number analyzed (Participants) | 7 | 2
Months | 7.5 [6.1 to 7.8] | NA [3.4 to NA] — Median was not estimable as data was available for only 1 participant and second participant was censored.

4. Secondary Outcome: Progression-Free Survival - Independent Review
Description: The below table shows Kaplan-Meier estimate of the median time from randomization to death from any cause or first observed disease progression.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trabectedin 1.5 mg/m2 | Trabectedin 0.58 mg/m2
Number analyzed (Participants) | 136 | 134
months | 3.3 [2.1 to 4.6] | 2.3 [2.0 to 3.4]
Statistical Analysis 1: Comparison: Trabectedin 1.5 mg/m2 vs Trabectedin 0.58 mg/m2; Test type: Superiority or Other; p = 0.0418, Log Rank; Hazard Ratio (HR) = 0.755, 95% CI 2-sided [0.574 to 0.992]

5. Secondary Outcome: Overall Survival
Description: as for outcome 4
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trabectedin 1.5 mg/m2 | Trabectedin 0.58 mg/m2
Number analyzed (Participants) | 136 | 134
months | 13.9 [12.5 to 18.6] | 11.8 [9.9 to 14.9]
Statistical Analysis 1: Comparison: Trabectedin 1.5 mg/m2 vs Trabectedin 0.58 mg/m2; Test type: Superiority or Other; p = 0.1920, Log Rank; Hazard Ratio (HR) = 0.843, 95% CI 2-sided [0.653 to 1.090]

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Trabectedin 1.5 mg/m2 | Trabectedin 0.58 mg/m2
Serious Adverse Events (participants affected / at risk) | 48/130 | 41/130
Other Adverse Events (participants affected / at risk) | 129/130 | 128/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trabectedin 1.5 mg/m2 (N=130) | Trabectedin 0.58 mg/m2 (N=130)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 2 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 1 | 3
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0
Mitral Valve Incompetence (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular Tachycardia (Cardiac disorders) | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 7 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 1 | 2
Small Intestinal Obstruction (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 3 | 2
Chest Discomfort (General disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Extravasation (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 0 | 1
Organ Failure (General disorders) | 0 | 1
Pain (General disorders) | 3 | 2
Pyrexia (General disorders) | 5 | 5
Arthritis Bacterial (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Catheter Related Infection (Infections and infestations) | 2 | 0
Empyema (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Perineal Abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 6 | 2
Sepsis (Infections and infestations) | 1 | 2
Septic Shock (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Wound Infection (Infections and infestations) | 0 | 1
Patella Fracture (Injury, poisoning and procedural complications) | 0 | 1
Radiation Pneumonitis (Injury, poisoning and procedural complications) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 0
Blood Bilirubin Increased (Investigations) | 1 | 0
Blood Creatinine Increased (Investigations) | 2 | 0
Blood Urea Increased (Investigations) | 1 | 0
Mediastinoscopy (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Liposarcoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour Associated Fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0
Depressed Level of Consciousness (Nervous system disorders) | 0 | 1
Nerve Compression (Nervous system disorders) | 0 | 1
Neuropathy (Nervous system disorders) | 0 | 1
Paresis (Nervous system disorders) | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 0 | 3
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Suicide Attempt (Psychiatric disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Non-Cardiogenic Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Abdominal Operation (Surgical and medical procedures) | 1 | 0
Bladder Catheterisation (Surgical and medical procedures) | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 1 | 0
Hepatectomy (Surgical and medical procedures) | 0 | 1
Hepatic Embolisation (Surgical and medical procedures) | 1 | 0
Laparotomy (Surgical and medical procedures) | 0 | 1
Lung Operation (Surgical and medical procedures) | 0 | 1
Mass Excision (Surgical and medical procedures) | 0 | 1
Sarcoma Excision (Surgical and medical procedures) | 2 | 0
Spinal Laminectomy (Surgical and medical procedures) | 1 | 0
Therapeutic Embolisation (Surgical and medical procedures) | 1 | 0
Tumour Excision (Surgical and medical procedures) | 1 | 0
Vitrectomy (Surgical and medical procedures) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 5 | 0
Embolism (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Shock (Vascular disorders) | 1 | 0
Thrombophlebitis Superficial (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trabectedin 1.5 mg/m2 (N=130) | Trabectedin 0.58 mg/m2 (N=130)
Anaemia (Blood and lymphatic system disorders) | 42 | 40
Leukopenia (Blood and lymphatic system disorders) | 16 | 9
Neutropenia (Blood and lymphatic system disorders) | 64 | 36
Thrombocytopenia (Blood and lymphatic system disorders) | 25 | 10
Abdominal Distension (Gastrointestinal disorders) | 8 | 10
Abdominal Pain (Gastrointestinal disorders) | 17 | 26
Abdominal Pain Upper (Gastrointestinal disorders) | 8 | 4
Constipation (Gastrointestinal disorders) | 45 | 45
Diarrhoea (Gastrointestinal disorders) | 30 | 28
Dyspepsia (Gastrointestinal disorders) | 8 | 12
Nausea (Gastrointestinal disorders) | 97 | 71
Vomiting (Gastrointestinal disorders) | 56 | 34
Asthenia (General disorders) | 26 | 26
Chest Pain (General disorders) | 6 | 15
Chills (General disorders) | 8 | 5
Fatigue (General disorders) | 76 | 72
Oedema (General disorders) | 4 | 7
Oedema Peripheral (General disorders) | 17 | 19
Pain (General disorders) | 8 | 11
Pyrexia (General disorders) | 31 | 18
Upper Respiratory Tract Infection (Infections and infestations) | 16 | 11
Alanine Aminotransferase Increased (Investigations) | 71 | 54
Aspartate Aminotransferase Increased (Investigations) | 62 | 38
Blood Alkaline Phosphatase Increased (Investigations) | 39 | 37
Blood Bilirubin Increased (Investigations) | 14 | 7
Blood Creatine Phosphokinase Increased (Investigations) | 14 | 19
Blood Creatinine Increased (Investigations) | 9 | 6
Haemoglobin Decreased (Investigations) | 9 | 8
Neutrophil Count Decreased (Investigations) | 16 | 5
Platelet Count Decreased (Investigations) | 7 | 4
Transaminases Increased (Investigations) | 7 | 2
Weight Decreased (Investigations) | 6 | 8
White Blood Cell Count Decreased (Investigations) | 11 | 8
Anorexia (Metabolism and nutrition disorders) | 29 | 21
Decreased Appetite (Metabolism and nutrition disorders) | 11 | 9
Dehydration (Metabolism and nutrition disorders) | 9 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 | 9
Hypocalcaemia (Metabolism and nutrition disorders) | 11 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 13 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 16
Back Pain (Musculoskeletal and connective tissue disorders) | 18 | 25
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 6 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 17 | 15
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 13 | 15
Dizziness (Nervous system disorders) | 18 | 14
Dysgeusia (Nervous system disorders) | 13 | 8
Headache (Nervous system disorders) | 37 | 35
Hypoaesthesia (Nervous system disorders) | 8 | 6
Paraesthesia (Nervous system disorders) | 9 | 6
Anxiety (Psychiatric disorders) | 11 | 9
Depression (Psychiatric disorders) | 9 | 9
Insomnia (Psychiatric disorders) | 20 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 34
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 3
Rash (Skin and subcutaneous tissue disorders) | 7 | 3
Hypotension (Vascular disorders) | 13 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days